CLINICAL TRIAL: NCT03287219
Title: Colon Staining Efficacy of Single Oral Doses of Methylene Blue MMX® Modified Release Tablets Administered to Patients Undergoing Colonoscopy
Brief Title: Colon Staining Efficacy of Single Oral Doses of Methylene Blue MMX
Acronym: CRO-11-108
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cosmo Technologies Ltd (Industry)
Collaborators: Cross S.A. (Industry)
Responsible Party: Sponsor
Organization: Cosmo Pharmaceuticals NV (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CB-17-01/03
Record Dates: First submitted 2017-08-22; First posted 2017-09-19 (Actual); Results first posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Colon Staining in Preparation for Colonoscopy

STUDY DESIGN:
Intervention Model Description: Open label, staining efficacy exploratory study.
Masking Description: None. Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 150 mg Methylene Blue-MMX tablets (Active Comparator): take 6 x 25mg Methylene Blue-MMX tablets equivalent to 150 mg
  Interventions: Drug: Methylene Blue MMX 25 mg modified release tablets
- 200 mg Methylene Blue-MMX tablets (Active Comparator): take 8 x 25mg Methylene Blue-MMX tablets equivalent to 200 mg
  Interventions: Drug: Methylene Blue MMX 25 mg modified release tablets

INTERVENTIONS:
Drug: Methylene Blue MMX 25 mg modified release tablets — Methylene Blue MMX 25 mg modified release tablets administered with a full dose regimen of a 4-L PEG-based bowel cleansing preparation.

SUMMARY:
To describe and evaluate the mucosal staining efficacy of Methylene Blue MMX® tablets after total oral doses of 150 or 200 mg in patients undergoing a full colonoscopy for various reasons.

DETAILED DESCRIPTION:
Objectives:

To describe and evaluate the mucosal staining efficacy of Methylene Blue MMX® tablets after total oral doses of 150 or 200 mg in patients undergoing a full colonoscopy for various reasons.

Primary end-point(s):

To evaluate the mucosal staining efficacy of Methylene Blue MMX® tablets after total oral doses of 150 or 200 mg.

Secondary end-point(s):

Bowel cleansing quality evaluated according to the validated Boston Bowel Preparation Scale (BBPS) after intake of 150 or 200 mg of Methylene Blue MMX® tablets during the intake of the bowel cleansing preparation.

To collect data about safety and tolerability of Methylene Blue MMX® tablets after administration of single oral doses of 150 or 200 mg.

Methodology:

Open label, staining efficacy exploratory study.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: males and females;
2. Age:18 to 70 years;
3. Colonoscopy: out-patients with indication for colonoscopy including faecal occult blood test positive colorectal cancer screening, polypectomy follow-up and inflammatory bowel disease check;
4. Contraception: either sterile subjects or subjects practising at least one reliable methods of contraception or in post-menopausal status for at least 1 year;
5. Informed Consent: signed written informed consent prior to inclusion in the study.

Exclusion Criteria:

1. Pregnancy: pregnant or lactating women or at a risk of becoming pregnant;
2. Allergy: known or suspected hypersensitivity to the active principle and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general;
3. Diseases: known or suspected gastrointestinal obstruction or perforation, toxic megacolon, major colonic resection, inflammatory bowel diseases in active phase, severe diverticulosis with diverticulitis, heart failure (Class III or IV), serious cardiovascular disease, severe liver failure, end-stage renal insufficiency, any other relevant disease that might interfere with the aim of the study.
4. Comprehension: inability to comprehend the full nature and purpose of the study and unwillingness to co-operate with the Investigator and to comply with the requirements of the entire study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2011-05-02 (Actual); Primary Completion 2012-01-16 (Actual); Study Completion 2012-01-16 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 150 mg Methylene Blue-MMX Tablets | 200 mg Methylene Blue-MMX Tablets
Started | 24 | 90
Completed | 24 | 88
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Methylene Blue MMX 150mg: Patients under going Colonoscpy taking Methylene Blue-MMX tablets equivalent to 150 mg
- Methylene Blue MMX 200mg: Patients under going Colonoscpy taking Methylene Blue-MMX tablets equivalent to 200 mg
- Total: Total of all reporting groups
Arm/Group | Methylene Blue MMX 150mg | Methylene Blue MMX 200mg | Total
Number analyzed (Participants) | 24 | 88 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (11.0) | 55.6 (11.2) | 54.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 35 | 46
  Male | 13 | 53 | 66
Height [Mean (Standard Deviation); unit: Centimetres] | 166.5 (8.4) | 168.5 (8.7) | 167.4 (8.7)
Body Weight [Mean (Standard Deviation); unit: Kg] | 68 (13.3) | 70.6 (14.2) | 69 (14.0)

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Mucosal Staining Efficacy
Description: Mucosal staining efficacy of Methylene Blue MMX tablets after total oral doses of 150 or 200 mg.
  Methylene blue staining efficacy was assessed by scoring the observed percentage of staining as reported below for each colon region (AC, TC, DC, RES) 0 - no staining
  1. - traces (poor traces in colon mucosa)
  2. - detectable (at least the 25% of colon mucosa is stained)
  3. - acceptable (at least the 50% of colon mucosa is stained)
  4. - good (at least the 75% of colon mucosa is stained)
  5. - over stained ( the 100% of the colon mucosa is over stained) After scoring (SC) separately each colonic segment, the total staining score (TSC) was also calculated and the number of regions with an SC>2 (NSA) was determined.
  For each patient, the best effective TSC was set at 16, when SC=4 was detected in all 4 regions. SC=5 detected in any region and TSC>16, both denoting an overstaining of the mucosa, were defined as suboptimal results in colon staining.
Time Frame: One day- mucosal staining efficacy is assessed during the colonoscopy procedure
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- A (Dose:150mg): Number of tablets taken in relation to the intake of the bowel cleansing preparation:
  At the beginning - 2 After the 1st L - 2 After the 2nd L - 2 After the 3rd L - 0 At the end - 0
- B (Dose:150mg): Number of tablets taken in relation to the intake of the bowel cleansing preparation:
  At the beginning - 6 After the 1st L - 0 After the 2nd L- 0 After the 3rd L- 0 At the end- 0
- C (Dose:150mg): Number of tablets taken in relation to the intake of the bowel cleansing preparation:
  At the beginning - 0 After the 1st L - 0 After the 2nd L - 0 After the 3rd L - 0 At the end - 6
- D (Dose:200mg); G (Dose 200mg): Number of tablets taken in relation to the intake of the bowel cleansing preparation At the beginning -4 After the 1st L-2 After the 2nd L-2 After the 3rd L-0 At the end-0
- E (Dose:200mg): Number of tablets taken in relation to the intake of the bowel cleansing preparation At the beginning -0 After the 1st L-0 After the 2nd L-0 After the 3rd L-0 At the end-8
- F (Dose:200mg): Number of tablets taken in relation to the intake of the bowel cleansing preparation At the beginning -2 After the 1st L-2 After the 2nd L-2 After the 3rd L-0 At the end-2
- H (Dose:200mg): Number of tablets taken in relation to the intake of the bowel cleansing preparation At the beginning -0 After the 1st L-0 After the 2nd L-0 After the 3rd L-4 At the end-4
- I (Dose:200mg): Number of tablets taken in relation to the intake of the bowel cleansing preparation At the beginning -0 After the 1st L-0 After the 2nd L-4 After the 3rd L-4 At the end-0
- J (Dose:200mg): Number of tablets taken in relation to the intake of the bowel cleansing preparation:
  At the beginning - 0 After the 1st L - 0 After the 2nd L - 2 After the 3rd L - 3 At the end - 3
Arm/Group | A (Dose:150mg) | B (Dose:150mg) | C (Dose:150mg) | D (Dose:200mg) | E (Dose:200mg) | F (Dose:200mg) | G (Dose 200mg) | H (Dose:200mg) | I (Dose:200mg) | J (Dose:200mg)
Number analyzed (Participants) | 8 | 7 | 9 | 20 | 9 | 8 | 2 | 20 | 16 | 13
scores on a scale | 6.8 (4.0) | 2.3 (2.4) | 8.1 (3.6) | 7.0 (5.0) | 9.8 (4.1) | 10.5 (4.1) | 10.5 (7.8) | 10.0 (3.2) | 11.4 (3.8) | 11.6 (3.5)

2. Secondary Outcome: Safety and Tolerability of Methylene Blue MMX as Determined by Vital Signs (Blood Pressure)
Description: safety and tolerability of Methylene Blue MMX reviewed by incidence of treatment emergent by measurement of vital signs (blood pressure)
Time Frame: until study completion (until 2 days after dose)
Population: Safety population: the safety population was defined as all enrolled subjects who received at least one dose of the study drug. This population was used for safety evaluation
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Pre Colonoscopy - 150mg Dose: Vital Signs - safety Population -- 150mg dose
- Pre Colonoscopy- 200mg Dose; During Colonoscopy- 200mg Dose; Post Colonoscopy- 200mg Dose: Vital Signs - safety Population- 200mg dose
- During Colonoscopy- 150mg Dose; Post Colonoscopy- 150mg Dose: Vital Signs - safety Population- 150mg dose
Arm/Group | Pre Colonoscopy - 150mg Dose | Pre Colonoscopy- 200mg Dose | During Colonoscopy- 150mg Dose | During Colonoscopy- 200mg Dose | Post Colonoscopy- 150mg Dose | Post Colonoscopy- 200mg Dose
Number analyzed (Participants) | 24 | 88 | 24 | 86 | 24 | 87
mmHg
  Systolic Blood Pressure (mmHg) | 122.6 (14.6) | 124.3 (17.7) | 122.6 (14.6) | 124.3 (17.7) | 122.7 (14.5) | 124.2 (17.7)
  Diastolic Blood Pressure(mmHg) | 74.7 (8.1) | 74.0 (11.9) | 74.9 (8.2) | 74.0 (11.9) | 75 (8.2) | 74.0 (11.9)

3. Secondary Outcome: Safety and Tolerability of Methylene Blue MMX as Determined by AEs
Description: Safety and tolerability of Methylene Blue MMX® tablets after administration of total oral doses of 150 or 200 mg.AEs were assessed throughout the study.
Time Frame: Until study completion (until 2 days after dose)
Measure: Count of Participants; unit: Participants
Arm/Group | Pre Colonoscopy - 150mg Dose | Pre Colonoscopy- 200mg Dose | During Colonoscopy- 150mg Dose | During Colonoscopy- 200mg Dose | Post Colonoscopy- 150mg Dose | Post Colonoscopy- 200mg Dose
Number analyzed (Participants) | 24 | 88 | 24 | 86 | 24 | 87
Participants | 3 | 3 | 0 | 0 | 0 | 0

4. Secondary Outcome: Safety and Tolerability of Methylene Blue MMX as Determined by Heart Rate
Description: incidence of treatment emergent by measurement of vital signs (heart rate) to determine Safety and Tolerability of Methylene Blue MMX
Time Frame: until study completion (until 2 days after dose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats per minute (BPM)
Groups:
- Pre Colonoscopy - 150mg Dose; During Colonoscopy - 150mg Dose; Post Colonoscopy- 150mg Dose: Vital Signs - safety Population - 150mg dose
- Pre Colonoscopy- 200mg Dose; During Colonoscopy- 200mg Dose; Post Colonoscopy- 200mg Dose: Vital Signs - safety Population - 200mg dose
Arm/Group | Pre Colonoscopy - 150mg Dose | Pre Colonoscopy- 200mg Dose | During Colonoscopy - 150mg Dose | During Colonoscopy- 200mg Dose | Post Colonoscopy- 150mg Dose | Post Colonoscopy- 200mg Dose
Number analyzed (Participants) | 24 | 87 | 24 | 85 | 24 | 87
beats per minute (BPM) | 73.9 (10.6) | 75.2 (15.1) | 74.3 (10.9) | 75.3 (15.1) | 74.2 (10.9) | 7.1 (15.1)

5. Secondary Outcome: Safety and Tolerability of Methylene Blue MMX as Determined by Vital Signs (Oxygen Saturation in Peripheral Blood)
Description: safety and tolerability of Methylene Blue MMX reviewed by incidence of treatment emergent by measurement of vital signs (Oxygen Saturation in peripheral blood)
Time Frame: until study completion (until 2 days after dose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of saturation
Groups:
- Pre Colonoscopy - 150mg Dose; During Colonoscopy- 150mg Dose; Post Colonoscopy- 150mg Dose: Vital Signs - safety Population
Arm/Group | Pre Colonoscopy - 150mg Dose | Pre Colonoscopy- 200mg Dose | During Colonoscopy- 150mg Dose | During Colonoscopy- 200mg Dose | Post Colonoscopy- 150mg Dose | Post Colonoscopy- 200mg Dose
Number analyzed (Participants) | 24 | 88 | 24 | 86 | 24 | 87
percentage of saturation | 98.4 (1.8) | 98.7 (6.6) | 98.4 (1.8) | 98.8 (6.5) | 98.4 (1.8) | 98.8 (6.5)

6. Secondary Outcome: Safety and Tolerability of Methylene Blue MMX as Determined Body Weight.
Description: safety and tolerability of Methylene Blue MMX in relation to incidence of treatment emergent by body weight.
Time Frame: until study completion (until 2 days after dose)
Measure: Mean (Standard Deviation); unit: Kg
Groups:
- Visit 1-Screening 150mL; Visit 2-Final 150mL: Safety Population 150mL Dose
- Visit 1-Screening 200mL; Visit 2-Final 200mL: Safety Population 200mL Dose
Arm/Group | Visit 1-Screening 150mL | Visit 1-Screening 200mL | Visit 2-Final 150mL | Visit 2-Final 200mL
Number analyzed (Participants) | 24 | 89 | 24 | 89
Kg | 67.2 (13.0) | 71.3 (15.9) | 67.4 (13.0) | 71.2 (15.8)

7. Secondary Outcome: Bowel Cleansing Quality-Boston Bowel Preparation Score
Description: Bowel cleansing quality evaluated according to the validated Boston Bowel Preparation Scale (BBPS).
  Colon was divided into 4 target regions: ascending colon (AC), transverse colon (TC), descending colon (DC) and rectosigmoid (RES). Methylene blue staining efficacy was assessed scoring the observed staining percentage as reported below for each colon region:
  0 - no staining
  1. - traces (poor traces in colon mucosa)
  2. - detectable (at least the 25% of colon mucosa is stained)
  3. - acceptable (at least the 50% of colon mucosa is stained)
  4. - good (at least the 75% of colon mucosa is stained)
  5. - over stained ( the 100% of the colon mucosa is over stained)
Time Frame: One day- bowel cleansing quality is assessed during the colonoscopy procedure
Measure: Mean (Standard Deviation); unit: Colon cleansing score
Groups:
- Overall: Overall Colon cleansing score
Arm/Group | 150 mg Methylene Blue-MMX Tablets | 200 mg Methylene Blue-MMX Tablets | Overall
Number analyzed (Participants) | 24 | 88 | 112
Colon cleansing score | 5.4 (1.7) | 5.4 (1.1) | 5.4 (1.2)

ADVERSE EVENTS:
Groups:
- AEs Methylene Blue-MMX Tablets Equivalent to 150 mg: Patients under going Colonoscpy taking Methylene Blue MMX Dose 150mL
- AEs Methylene Blue-MMX Tablets Equivalent to 200 mg: Patients under going Colonoscpy taking Methylene Blue MMX dose 200 mg
Arm/Group | AEs Methylene Blue-MMX Tablets Equivalent to 150 mg | AEs Methylene Blue-MMX Tablets Equivalent to 200 mg
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/88
Other Adverse Events (participants affected / at risk) | 1/24 | 2/88
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AEs Methylene Blue-MMX Tablets Equivalent to 150 mg (N=24) | AEs Methylene Blue-MMX Tablets Equivalent to 200 mg (N=88)
vomiting (Gastrointestinal disorders) | 1 (3) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes